CLINICAL TRIAL: NCT06485063
Title: Effects of Myofascial Reorganization on Running Performance, and Lower Limb Biomechanical, Viscoelastic, and Thermographic Properties of Triathletes: a Randomized Clinical Trial.
Brief Title: Myofascial Reorganization on Performance, and Biomechanical, Viscoelastic, and Thermographic Properties of Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Principal Investigator, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Performance in athletes
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: athletes; performance; healthy; fascia

STUDY DESIGN:
Intervention Model Description: Two-arm Randomized Clinical Trial, presenting a placebo and a experimental group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to which group they will belong, as they never had contact to the technique investigated. The statistical analysis will be blinded as well, and the statistical will not know which is the experimental or the placebo group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Reorganization Group (Experimental): Each participant will receive 12 sessions of Myofascial Reorganization
  Interventions: Other: Myofascial Reorganization
- Placebo Myofascial Reorganization (Placebo Comparator): Each participant will receive 12 sessions of Myofascial Reorganization Placebo
  Interventions: Other: PLACEBO Myofascial Reorganization

INTERVENTIONS:
Other: Myofascial Reorganization — It is a manual technique in which the therapist applies a manual sustained oblique load of 45° with subsequent shear load. In general, the technique is divided into two stages, the first when the oblique load is accompanied by a passive shear load (applied by the therapist) during 1minute, and the second stage, when the shear oblique manual load is maintained but the shear load provoked by the participants' active movement (active shear load) during 1minute.
  Other Names: RMF; Reorganização Miofascial
  Arms: Myofascial Reorganization Group
Other: PLACEBO Myofascial Reorganization — it is light touch to the skin applied by the therapist, without provoking compression, or any constant or shear load during the fist minute. In the second minute, the participant adds active movements to the light touch. This two stage (each one during 1minute) is constructed to mimic the passive and the active stages of the real myofascial reorganization technique.
  Other Names: RMF-PLACEBO; Reorganização Miofascial Placebo
  Arms: Placebo Myofascial Reorganization

SUMMARY:
This is a two-group randomized clinical trial (includes an experimental and a placebo group) to verify the effects of the Myofascial Reorganization (RMF) compared to the placebo-RMF technique on running performance and thermographic, biomechanical, and viscoelastic proprieties of lower limbs of male triathletes. Data collection will be carried out one week before the first intervention session, and one week after the last intervention session. Anthropometric characteristics (height and weight), lower limbs, and biomechanical, viscoelastic, and thermographic properties will be collected before any exercise tests. After this, the athlete will be submitted to: a 10-minute protocol to verify running economy on the treadmill, followed by an incremental test on the treadmill, and a time to exhaustion test. Evaluation procedures will carried out one week before (0 weeks) and one week after (7th week) the experimental/placebo intervention. Intervention sessions will occur during six weeks, twice a week, each session lasting up to 30 minutes.

DETAILED DESCRIPTION:
1. This study was approved by the Ethical Committee involving Research with Human Beings of the University of Santa Catarina (UDESC) under protocol number 56498722.1.0000.0118. Consolidated Standards of Reporting Trials will be followed.

2.1 General objectives: to verify the effects of the Myofascial Reorganization (RMF) technique compared to the placebo-RMF technique on running performance and thermographic, biomechanical, and viscoelastic proprieties of lower limbs of athletes.

2.2 Specific objectives: intragroup and intergroup comparisons of running-related performance variables, lower limb skin temperature, and biomechanical and viscoelastic properties.

3. Sample: Athletes volunteers living in Florianópolis, SC, Brazil, if they meet inclusion criteria and do not meet exclusion criteria.

4. Sampling: will be non-probabilistic by convenience and snowball (participants will be recruited by social media, flyers, and by referral of other participants).

5. Data collection procedures: the athletes will be evaluated before (0 weeks) and after (7 weeks) a 6-week intervention protocol.

5.1 Anthropometric measures: height (centimeters) will be collected using a stadiometer, and body mass (kilograms) will be measured using a weighting balance.

5.2 Lower limb skin temperature: Thermographic characteristics of lower limbs will be measured in a dark and controlled room, at an ambient temperature of 24°C(±1°) and relative air humidity of 50%, after 15 minutes of acclimatation. Anterior and posterior lower limb regions of interest will be included.

5.3 Biomechanical and viscoelastic properties:

Biomechanical and viscoelastic properties State of tension, biomechanical and viscoelastic properties of the myofascial tissue of lower limbs and thoracolumbar region will be assessed using a non-invasive digital palpation device. These properties will be:

* F: Frequency
* S: Dynamic Stiffness
* D: logarithmic decrement
* R: Relaxation time,
* C: Creep. These measures will be taken bilaterally on the anterior and posterior regions of the tights, the iliotibial tract, and the thoracolumbar region.

5.4 Performance-related tests: all exercise tests to analyze running performance-related variables will be carried out on a treadmill while monitoring the heart rate using a frequency meter and analyzing the gas exchange parameters using a gas analyzer in an open circuit breath-by-breath.

5.4.1 Running Economy: is the oxygen consumption at a common velocity, chosen to be under the first lactate threshold. The athletes will run at a constant velocity of 7 kilometers per hour while measuring their oxygen consumption (VO2) and monitoring the heart rate, for 10 minutes.

5.4.3 Incremental 3-minute graded test: The maximal volume of oxygen consumption (VO2 max), the maximal velocity of the incremental test, and lactate thresholds will be determined by an incremental graded test until volitional exhaustion, using stages of 3min, and an increment of 1km/h per stage, with a slope of 1% on the treadmill. Between each stage, capillary blood from the ear lobe will be collected to determine lactate blood concentrations. The perceived effort will be measured using the 10-point scale for perceived effort.

5.4.4 Lactate thresholds: blood lactate concentrations [bLa] will be derived from blood samples collected from the ear lobe during the incremental test, and the first (LT1) and the second lactate threshold (LT2) will be determined.

5.4.5 Time to Exhaustion Test: to determine the time to exhaustion in a maximal effort and as a verification of the VO2max. After the 20-minute rest after the incremental test, a re-warm of 3 minutes will be taken at a velocity of 50% of the maximal velocity reached by the incremental test. Then, the athlete will perform the test at 100% of the maximal velocity, until volitional exhaustion.

6 Groups and Interventions

After an evaluation (0 weeks), the participants will be randomized into one of the two groups: (a) Myofascial Reorganization (RMF) or (b) PLACEBO Myofascial Reorganization (RMFplacebo). They will be blinded to the group of intervention. The randomization will be enrolled using sealed envelopes, and the allocation will be carried out in blocks of 4 by a non-investigator.Both groups will receive 6 weeks of experimental/placebo intervention, twice a week. Each session will last approximately 30 minutes. The RMF group will receive a specific mechanical load directed to the fascial system (real technique) while the placebo group will receive a simulation of the technique (a light touch to the skin), added to lower limb voluntary movements. The real technique consists of a specific 45° oblique mechanical load applied to the fascial system, and it includes an additional shear load provoked passively (by the therapist) and then actively (provoked by the participant's voluntary movement).The re-tests will be carried out one week after the last session of intervention (in the 7th week).RMF will be applied:

6.1. Thoracolumbar fascia insertion: using one proximal hand (closer to the participant's head) and a distal hand (closer to the participant's feet). Proximal hand - three fingers on the iliolumbar ligament. Distal hand - three fingers on the lateral edge of the sacrum. Passive load (first stage): the therapist applies a progressive then sustained oblique 45° load with both hands, directing the force vector to the pelvis center, with additional craniocaudal shear load, using the fingers, both hands working synchronically. Active load (second stage): the participant, lying in the supine position, contralateral and ipsilateral lower limbs initially relaxed, both feet placed in the stretcher and hips, and knees flexed at 90°/90°, hands on the thorax, starts, with ipsilateral lower limb will perform an active movement: (a) hip external rotation, added to dorsal flexion of the ankle, and flexion of the knee, and hip joints; (b) followed by the movement of hip internal rotation added to plantar flexion of the ankle, and extension knee, and hip joints.

6.2. Abdominal muscles fascia: The therapist's hands are placed on a virtual triangle formed by the anterior iliac spine, the umbilical scar, and the pubic symphysis, closer to the insertion of the abdominis muscles on the pelvis, where the fascia of rectus abdominis muscle and the obliques muscles separate. First stage: the therapist's fingers will be directed to the center of the pelvis, the hands working synchronically. The therapist applies a progressive mechanical oblique load directing the force vector to the pelvis center, adding a subsequent shear load in the craniocaudal direction, with both hands working synchronically. The participant lies on the stretcher in supine, contralateral, and ipsilateral lower limbs initially relaxed, both feet placed in the stretcher, hips, and knees flexed at 90°/90°, and the hands on the thorax. In the second stage, the participant will add ante/retroversion of the pelvis to promote the active shear load.

6.3. Quadriceps femoris muscle: The therapist will use a proximal and a distal hand. Proximal hand: acting as an anchor - the hypothenar region in parallel with the lateral side of the participant, contemplating the surface between both anterior and inferior iliac spines; to perform that anchor, the therapist will bring the skin excess and apply a soft and sustained mechanical load until they find the fascial barrier. Distal hand: the therapist's hand will embrace the distal portion of the tight, contemplating the patella, the first finger on the lateral side of the knee region, and the other fingers on the medial side; the fingers will create an anchor, promoting an "intention" to separate the quadriceps femoris muscle from the iliotibial tract and the insertion of the sartorius, gracious and semitendinosus muscles. At the same time, using these fingers, the caudal hand will apply the mechanical load with the subsequent shear load. First stage: the mechanical oblique load is applied with a subsequent shear load in the proximal-distal direction. Second stage: passive shear load is replaced by the active shear load (movement with the ipsilateral lower limb). The participant will be in the supine position. The ipsilateral lower limb lies on the therapist's tight (that acts as a cushion, under the knee region), knee flexed between 40° and 50°, foot resting on the stretcher. The contralateral lower limb: foot resting on the stretcher, keeping 90°/90° hip and knee flexion. The ipsilateral will perform, slowly and with a short range of motion, cycles of knee flexion added to dorsiflexion, followed by knee extension and plantar flexion. The cycle is repeated during the stage time.

6.4. a. Fascia lata tensor muscle and iliotibial tract: the therapist will place one hand right beside the other, with the thumbs relaxed, and the other fingers semi-flexed as if the hands formed a "C". The hands will mirror each other, the carpi bones of the right hand almost touching the ones of the left hand. Both hands will be placed on the supra-trochanteric region. Stage one: The load will be applied using the hypothenar region of the right and left hands and the lateral surface of the 5th right and left fingers. The mechanical oblique load will be directed to the center of the pelvis and knee, with a passive shear load in the mediolateral direction. Stage two: the participant will be in lateral decubitus, relaxed, with the ipsilateral hip in light flexion, the knee in extension, and the contralateral lower limb with hip and knee flexed at 90°/90°. The ipsilateral lower limb executes a hip and knee flexion added to ankle dorsal flexion, then a hip and knee extension added to an ankle plantar flexion, repeatedly.

6.4. b. Fascia lata tensor muscle and iliotibial tract: the therapist will use a medial hand (placed on the medial side of the knee), acting as an anchor, and one lateral hand (lateral side of the knee), that will apply the mechanical load. Anchor (medial hand): the thumb embraces medial the region of the knee. Mechanical load (lateral hand): on the lateral region of the tight, 5cm above the articular line, on the insertion of the iliotibial tract; the hypothenar region of the hand will apply the load 5cm above the joint line of the knee (the distal third of the iliotibial tract). Stage one: The lateral hand applies the mechanical oblique load, vector directed to the center of the pelvis, and to the ceiling, with the shear load applied in the mediolateral direction. Stage two: the participant, already in lateral decubitus, with the contralateral lower limb in 90/90° hip and knee flexion, and the ipsilateral initially, the hip in light flexion, and the knee in extension will perform a very short range of motion of hip internal rotation and then returns to the initial position, repeatedly, with the ipsilateral lower limb.

6.4. c. Fascia lata tensor muscle and iliotibial tract: from the abovementioned position, only the second stage (active shear load) is repeated, but the therapist's mechanical load hand (lateral hand) is now on the proximal insertion of the iliotibial tract.

6.5 Hamstrings muscles: The participant will be in the supine position, contralateral lower limb with the foot resting on the stretcher, keeping the hip and the knee flexed at 90°/90°. The participant's ipsilateral knee initially rested on the therapist's shoulder. The therapist uses one hand to stabilize the participant's knee, and the other hand, to promote the mechanical load. Stabilizing hand: on the distal region of the thigh, involving the knee and stabilizing the participant's limb. Mechanical load hand: the therapist will apply the mechanical load using the diaphysis of the distal phalanges; on the proximal third of the tight, close to the insertion of the ipsilateral hamstring muscles. Stage one: progressive then sustained 45° oblique load, force vector directed to the center of the pelvis added to a shear load in the proximal-distal direction (from the ischiatic bone to the knee, repeatedly). Stage two: the participant's ipsilateral lower limb performs knee flexion/extension (not full extension).

6.6 Adductor muscles: The participant will be in the supine position. The Ipsilateral lower limb with the foot resting on the stretcher, the tight resting against the therapist's tight, maintaining a hip and knee flexion of approximately 60°/60°, and slight hip external rotation. The contralateral lower limb with the foot resting in the stretcher, maintaining 90°/90° of hip and knee flexion. The therapist will use one hand as an anchor, while the other applies the mechanical load. Anchor: the thumb performs an oblique 45°load directed to the center of the pelvis, on the region that designs a virtual triangle formed by the umbilical scar, the anterior superior iliac spine, and the pubic symphysis. Hand of the mechanical load: performing thumb opponency while the second and third fingers remain together, in interphalangeal and metacarpophalangeal flexion, forming a "C", this hand promotes a continuous mechanical load, 15cm distant to the pubic symphysis. Stage one: progressive then sustained 45° oblique load, force vector directed to the center of the pelvis, with additional shear load on the proximal-distal direction (from the pelvis to the knee, and vice-versa). Stage two: the participant will perform, with the ipsilateral lower limb, hip internal/external rotation repeatedly.

The placebo technique will repeat all the stages, except the therapist will apply a light touch to the skin during stages one and two. The movements of stage two will be performed.

7Statistical Analysis The data will be processed using IBM Statistical Package for the Social Sciences version 20.0. The Shapiro-Wilk test will determine the normality of data, and an analysis of variance (ANOVA) 2x2 will be conducted to compare between conditions (experimental/placebo) and between the baseline (0 weeks) and post-intervention (7th week). All analyses will be bidirectional and set to a significance level of (p<0,05). The effect size will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Athletes
* Age between 18 and 45 years
* 2 years of competitive experience
* Non-smokers
* Training at least 3 times/week intending to compete in at least local competitions
* No presenting lower limb surgery in the last 12 months
* Not presenting lower limb injury in the last 6 months
* Not presenting cerebellar diseases that limit sportive practice
* Not presenting brain diseases that limit sportive practice
* Not presenting musculoskeletal diseases that limit sportive practice
* Not presenting signs of rhabdomyolysis
* Not presenting systemic conditions that limit sportive practice
* Not presenting metabolic that limits sports practice
* Not presenting autoimmune conditions;
* Not presenting cardiac conditions.

Exclusion Criteria:

* Not accomplishing 83,3% (10 of 12 sessions) of the proposed experimental/placebo protocol
* Not presenting themselves on the re-test day
* Developing a lower limb musculoskeletal injury during the study's ongoing period.
* Developing a back injury during the study's ongoing period?
* Developing central or peripheral nervous system conditions during the study's ongoing period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Running Economy | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  the volume consumption of oxygen (VO2) required at a common velocity under the first lactate threshold in milliliters per minute per kilogram (mL.min-1.Kg-1).
Maximal volume consumption of oxygen | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  The maximal volume consumption of oxygen (VO2max) in milliliters per minute per kilogram (mL.min-1.Kg-1) will be determined as the highest value reached in the last stage plotted employing means of 15 seconds.
Time to Exhaustion | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  Time to volitional exhaustion during the Time to Exhaustion Test, running at 100% of the last velocity reached in the incremental test, in minutes and seconds.
Maximal velocity | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  maximal velocity derived from the incremental graded test

SECONDARY OUTCOMES:
State of tension: F - Frequency or TONE | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  Frequency of natural oscillation in Hz, characterized as TONE or state of tension;
Dynamic Stiffness (N/m); | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  the force (in Nelton) required to deform a meter of area
D -logarithmic decrement | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  characterized as ELASTICITY or dissipation of the natural oscillation (arbitrary units);
R- Relaxation time | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  the time to relaxation after mechanical stress (ms)
C - Creep | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  or reason between the relaxation time and the oscillation time, or Deborah number (used to characterize the fluidity of the materials in specific conditions of flux
First lactate threshold | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  the point in the curve where the lactate concentration per liter of blood approximates the concentration of 2 mmol/L, counting from the baseline
Second lactate threshold | Pre-intervention (0 week time point) and post-intervention (7 week time point)
  determined as a point equivalent to the rise of 4 millimoles per liter (mmol/L) from the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Health and Sport Sciences of the State University of Santa Catarina, Florianópolis, Santa Catarina, Brazil

REFERENCES:
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Okano, A. H. et al. Comparação entre limiar anaeróbio determinado por variáveis ventilatórias e pela resposta do lactato sanguíneo em ciclistas. Rev. Bras. Med. do Esporte 12, 39-44 (2006).
- [Background] Borszcz, F. K. Reprodutibilidade e validade do functional threshold power em ciclistas. (Universidade do Estado de Santa Catarina, 2018).
- [Background] McKay AKA, Stellingwerff T, Smith ES, Martin DT, Mujika I, Goosey-Tolfrey VL, Sheppard J, Burke LM. Defining Training and Performance Caliber: A Participant Classification Framework. Int J Sports Physiol Perform. 2022 Feb 1;17(2):317-331. doi: 10.1123/ijspp.2021-0451. Epub 2022 Dec 29. PMID 34965513
- [Background] Moran RN, Hauth JM, Rabena R. The effect of massage on acceleration and sprint performance in track & field athletes. Complement Ther Clin Pract. 2018 Feb;30:1-5. doi: 10.1016/j.ctcp.2017.10.010. Epub 2017 Oct 28. PMID 29389467
- [Background] Healey KC, Hatfield DL, Blanpied P, Dorfman LR, Riebe D. The effects of myofascial release with foam rolling on performance. J Strength Cond Res. 2014 Jan;28(1):61-8. doi: 10.1519/JSC.0b013e3182956569. PMID 23588488
- [Background] Fletcher IM. The effects of precompetition massage on the kinematic parameters of 20-m sprint performance. J Strength Cond Res. 2010 May;24(5):1179-83. doi: 10.1519/JSC.0b013e3181ceec0f. PMID 20386129
- [Background] Dibai-Filho AV, Guirro EC, Ferreira VT, Brandino HE, Vaz MM, Guirro RR. Reliability of different methodologies of infrared image analysis of myofascial trigger points in the upper trapezius muscle. Braz J Phys Ther. 2015 Mar-Apr;19(2):122-8. doi: 10.1590/bjpt-rbf.2014.0076. Epub 2015 Apr 27. PMID 25993626
- [Background] Inglis EC, Iannetta D, Passfield L, Murias JM. Maximal Lactate Steady State Versus the 20-Minute Functional Threshold Power Test in Well-Trained Individuals: "Watts" the Big Deal? Int J Sports Physiol Perform. 2019 Nov 4;15(4):541-547. doi: 10.1123/ijspp.2019-0214. Print 2020 Apr 1. PMID 31689684
- [Background] Borszcz FK, Tramontin AF, Bossi AH, Carminatti LJ, Costa VP. Functional Threshold Power in Cyclists: Validity of the Concept and Physiological Responses. Int J Sports Med. 2018 Oct;39(10):737-742. doi: 10.1055/s-0044-101546. Epub 2018 May 25. PMID 29801189
- [Background] Corte AC, Pedrinelli A, Marttos A, Souza IFG, Grava J, Jose Hernandez A. Infrared thermography study as a complementary method of screening and prevention of muscle injuries: pilot study. BMJ Open Sport Exerc Med. 2019 Jan 3;5(1):e000431. doi: 10.1136/bmjsem-2018-000431. eCollection 2019. PMID 30687515
- [Background] Bravo-Sanchez A, Abian P, Sanchez-Infante J, Esteban-Gacia P, Jimenez F, Abian-Vicen J. Objective Assessment of Regional Stiffness in Vastus Lateralis with Different Measurement Methods: A Reliability Study. Sensors (Basel). 2021 May 6;21(9):3213. doi: 10.3390/s21093213. PMID 34066343
- [Background] Alaca N, Kablan N. Acute effects of cold spray application on mechanical properties of the rectus femoris muscle in athletes. J Bodyw Mov Ther. 2022 Apr;30:100-104. doi: 10.1016/j.jbmt.2022.02.010. Epub 2022 Feb 7. PMID 35500956
- [Background] Frohlich-Zwahlen AK, Casartelli NC, Item-Glatthorn JF, Maffiuletti NA. Validity of resting myotonometric assessment of lower extremity muscles in chronic stroke patients with limited hypertonia: a preliminary study. J Electromyogr Kinesiol. 2014 Oct;24(5):762-9. doi: 10.1016/j.jelekin.2014.06.007. Epub 2014 Jun 24. PMID 25023163
- [Background] Schoenrock B, Zander V, Dern S, Limper U, Mulder E, Veraksits A, Viir R, Kramer A, Stokes MJ, Salanova M, Peipsi A, Blottner D. Bed Rest, Exercise Countermeasure and Reconditioning Effects on the Human Resting Muscle Tone System. Front Physiol. 2018 Jul 3;9:810. doi: 10.3389/fphys.2018.00810. eCollection 2018. PMID 30018567
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Konrad, A. & Paternoster, F. K. No Association between Jump Parameters and Tissue Stiffness in the Quadriceps and Triceps Surae Muscles in Recreationally Active Young Adult Males. Appl. Sci. 12, (2022).
- [Background] Hill M, Rosicka K, Wdowski M. Effect of sex and fatigue on quiet standing and dynamic balance and lower extremity muscle stiffness. Eur J Appl Physiol. 2022 Jan;122(1):233-244. doi: 10.1007/s00421-021-04831-0. Epub 2021 Oct 20. PMID 34669045
- [Background] Hill MW, Wdowski MM, Rosicka K, Kay AD, Muehlbauer T. Exploring the relationship of static and dynamic balance with muscle mechanical properties of the lower limbs in healthy young adults. Front Physiol. 2023 May 26;14:1168314. doi: 10.3389/fphys.2023.1168314. eCollection 2023. PMID 37304823
- [Background] Bizzini M, Mannion AF. Reliability of a new, hand-held device for assessing skeletal muscle stiffness. Clin Biomech (Bristol). 2003 Jun;18(5):459-61. doi: 10.1016/s0268-0033(03)00042-1. PMID 12763442
- [Background] Langevin HM, Stevens-Tuttle D, Fox JR, Badger GJ, Bouffard NA, Krag MH, Wu J, Henry SM. Ultrasound evidence of altered lumbar connective tissue structure in human subjects with chronic low back pain. BMC Musculoskelet Disord. 2009 Dec 3;10:151. doi: 10.1186/1471-2474-10-151. PMID 19958536
- [Background] Barnes KR, Kilding AE. Running economy: measurement, norms, and determining factors. Sports Med Open. 2015 Dec;1(1):8. doi: 10.1186/s40798-015-0007-y. Epub 2015 Mar 27. PMID 27747844
- [Background] Paton CD, Hopkins WG. Combining explosive and high-resistance training improves performance in competitive cyclists. J Strength Cond Res. 2005 Nov;19(4):826-30. doi: 10.1519/R-16334.1. PMID 16287351
- [Background] Costa, V. P. Efeitos de um bloco semanal de treinamento intervalado de alta intensidade nos índices fisiológicos e performance de ciclistas competitivos. (Universidade Federal de Santa Catarina, 2014).
- [Background] Jamnick NA, Botella J, Pyne DB, Bishop DJ. Manipulating graded exercise test variables affects the validity of the lactate threshold and V ⁢ O 2 ⁢ peak . PLoS One. 2018 Jul 30;13(7):e0199794. doi: 10.1371/journal.pone.0199794. eCollection 2018. PMID 30059543
- [Background] Amann M, Subudhi A, Foster C. Influence of testing protocol on ventilatory thresholds and cycling performance. Med Sci Sports Exerc. 2004 Apr;36(4):613-22. doi: 10.1249/01.mss.0000122076.21804.10. PMID 15064589
- [Background] Rohrken G, Held S, Donath L. Six Weeks of Polarized Versus Moderate Intensity Distribution: A Pilot Intervention Study. Front Physiol. 2020 Nov 12;11:534688. doi: 10.3389/fphys.2020.534688. eCollection 2020. PMID 33281607
- [Background] De Pauw K, Roelands B, Cheung SS, de Geus B, Rietjens G, Meeusen R. Guidelines to classify subject groups in sport-science research. Int J Sports Physiol Perform. 2013 Mar;8(2):111-22. doi: 10.1123/ijspp.8.2.111. PMID 23428482
- [Background] Kuipers H, Rietjens G, Verstappen F, Schoenmakers H, Hofman G. Effects of stage duration in incremental running tests on physiological variables. Int J Sports Med. 2003 Oct;24(7):486-91. doi: 10.1055/s-2003-42020. PMID 12968205
- [Background] Mugele H, Plummer A, Baritello O, Towe M, Brecht P, Mayer F. Accuracy of training recommendations based on a treadmill multistage incremental exercise test. PLoS One. 2018 Oct 11;13(10):e0204696. doi: 10.1371/journal.pone.0204696. eCollection 2018. PMID 30307961
- [Background] Borg G. Psychophysical scaling with applications in physical work and the perception of exertion. Scand J Work Environ Health. 1990;16 Suppl 1:55-8. doi: 10.5271/sjweh.1815. PMID 2345867
- [Background] Possamai LT, Borszcz FK, de Aguiar RA, de Lucas RD, Turnes T. Agreement of maximal lactate steady state with critical power and physiological thresholds in rowing. Eur J Sport Sci. 2022 Mar;22(3):371-380. doi: 10.1080/17461391.2021.1874541. Epub 2021 Feb 8. PMID 33428539
- [Background] Schlickmann, J. Suplementação com bicarbonato de sódio: influência sobre o desempenho, respostas fisiológicas e neuromusculares durante e após o exercício supramáximo no ciclismo. (2012)
- [Background] Bentley DJ, McNaughton LR, Batterham AM. Prolonged stage duration during incremental cycle exercise: effects on the lactate threshold and onset of blood lactate accumulation. Eur J Appl Physiol. 2001 Aug;85(3-4):351-7. doi: 10.1007/s004210100452. PMID 11560091
- [Background] Binder RK, Wonisch M, Corra U, Cohen-Solal A, Vanhees L, Saner H, Schmid JP. Methodological approach to the first and second lactate threshold in incremental cardiopulmonary exercise testing. Eur J Cardiovasc Prev Rehabil. 2008 Dec;15(6):726-34. doi: 10.1097/HJR.0b013e328304fed4. PMID 19050438
- [Background] Asplund CA, O'Connor FG, Noakes TD. Exercise-associated collapse: an evidence-based review and primer for clinicians. Br J Sports Med. 2011 Nov;45(14):1157-62. doi: 10.1136/bjsports-2011-090378. Epub 2011 Sep 26. PMID 21948122
- [Background] Van Hooren B, Peake JM. Do We Need a Cool-Down After Exercise? A Narrative Review of the Psychophysiological Effects and the Effects on Performance, Injuries and the Long-Term Adaptive Response. Sports Med. 2018 Jul;48(7):1575-1595. doi: 10.1007/s40279-018-0916-2. PMID 29663142
- [Background] Anley C, Noakes T, Collins M, Schwellnus MP. A comparison of two treatment protocols in the management of exercise-associated postural hypotension: a randomised clinical trial. Br J Sports Med. 2011 Nov;45(14):1113-8. doi: 10.1136/bjsm.2010.071951. Epub 2010 Jun 28. PMID 20584756
- [Background] Ostrow CL. Use of the Trendelenburg position by critical care nurses: Trendelenburg survey. Am J Crit Care. 1997 May;6(3):172-6. PMID 9131195
- [Background] WHO Guidelines on Drawing Blood: Best Practices in Phlebotomy. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138650/ PMID 23741774
- [Background] Chen G, Wu J, Chen G, Lu Y, Ren W, Xu W, Xu X, Wu Z, Guan Y, Zheng Y, Qiu B. Reliability of a portable device for quantifying tone and stiffness of quadriceps femoris and patellar tendon at different knee flexion angles. PLoS One. 2019 Jul 31;14(7):e0220521. doi: 10.1371/journal.pone.0220521. eCollection 2019. PMID 31365582
- [Background] Christiansen L, Larsen MN, Madsen MJ, Grey MJ, Nielsen JB, Lundbye-Jensen J. Long-term motor skill training with individually adjusted progressive difficulty enhances learning and promotes corticospinal plasticity. Sci Rep. 2020 Sep 24;10(1):15588. doi: 10.1038/s41598-020-72139-8. PMID 32973251
- [Background] Jedrzejewski G, Kasper-Jedrzejewska M, Dolibog P, Szygula R, Schleip R, Halski T. The Rolf Method of Structural Integration on Fascial Tissue Stiffness, Elasticity, and Superficial Blood Perfusion in Healthy Individuals: The Prospective, Interventional Study. Front Physiol. 2020 Sep 15;11:1062. doi: 10.3389/fphys.2020.01062. eCollection 2020. PMID 33041843
- [Background] Dos Santos Amorim M, Sinhorim L, Wagner J, de Paula Lemos F, Schleip R, Sonza A, Santos GM. Acute effects of myofascial reorganization on trapezius muscle oxygenation in individuals with nonspecific neck pain. J Bodyw Mov Ther. 2022 Jan;29:286-290. doi: 10.1016/j.jbmt.2021.10.010. Epub 2021 Oct 21. PMID 35248284
- [Background] Franca MED, Sinhorim L, Martins DF, Schleip R, Machado-Pereira NAMM, de Souza GM, Horewicz VV, Santos GM. Manipulation of the Fascial System Applied During Acute Inflammation of the Connective Tissue of the Thoracolumbar Region Affects Transforming Growth Factor-beta1 and Interleukin-4 Levels: Experimental Study in Mice. Front Physiol. 2020 Dec 3;11:587373. doi: 10.3389/fphys.2020.587373. eCollection 2020. PMID 33424619
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Background] Cohen, J. Statistical Power Analysis for the Behavioral Sciences. (Lawrence Erlbaum Associates, 1988).